CLINICAL TRIAL: NCT00441272
Title: Pioglitazone for Hepatic Steatosis in HIV
Brief Title: Pioglitazone to Treat Fatty Liver in People With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Colleen M. Hadigan, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 070105; 07-I-0105
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2008-10

CONDITIONS: HIV Infections; Hepatic Steatosis; Insulin Resistance
Keywords: Pioglitazone; Hepatic Steatosis; Liver Toxicity; Liver Biopsy; HIV; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Fatty Liver; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
This study will determine whether pioglitazone (Actos, a drug approved to treat diabetes, can benefit HIV-infected people with fatty liver. Fatty changes of the liver (also known as steatosis) have been linked to diabetes and long-term liver damage in some patients. Pioglitazone has been shown to improve fatty liver in people without HIV; this study will see if it is beneficial for people with HIV as well.

HIV-infected patients 18 years of age and older with increased fat in the liver may be eligible for this study. Screening includes a CT scan and liver biopsy (withdrawal of a small sample of liver tissue through a needle).

Participants are randomly assigned to take either 45 mg of pioglitazone or placebo (sugar pill) by mouth once a day for 48 weeks. At the end of 48 weeks, all participants stop taking their medication and are followed for an additional 48 weeks to see what, if any benefits, of pioglitazone persist after treatment is stopped. In addition to taking the study medication, participants undergo the following procedures:

* Visits to the NIH Clinical Center over a period of approximately 2 years at day 0 and weeks 2, 8, 16, 24, 32, 40, 48, 52, 72, and 96. Most visits take about 1 hour and include blood drawing for various laboratory tests.
* Insulin clamp test at day 0 and weeks 24 and 48 to see how the body processes glucose. This test takes 4 to 6 hours and may include an overnight stay at the Clinical Center. A catheter (plastic tube) is placed in a vein in the arm to infuse insulin and another is placed in a vein on the back of the hand to draw blood samples. Blood sugar is checked frequently and glucose is given to keep blood sugar at normal values.
* Nutrition evaluations at day 0 and weeks 24 and 48. Subjects write down all the food they eat and drink for 4 days before the visit. They meet with a nutritionist to review the food record and to complete simple measurements of body fat and shape.
* CT scan of liver and abdomen at weeks 24, 48, 72 and 96.
* Liver biopsy at week 48.

DETAILED DESCRIPTION:
While the introduction of antiretroviral therapy for HIV/AIDS has transformed HIV disease into a chronic infection for many, the use of antiretroviral therapy is also often associated with metabolic abnormalities including insulin resistance, central fat accumulation and peripheral fat atrophy. Fatty infiltration of the liver or hepatic steatosis may be an important consequence of these metabolic derangements or may represent a direct toxicity associated with HIV infection and/or antiretroviral medications. Preliminary data suggests that hepatic steatosis may be very common and perhaps present in up to 50 percent of HIV-infected patients receiving antiretroviral therapy. Hepatic steatosis represents one step in the potential progression towards hepatocellular injury, non-alcoholic steatohepatitis (NASH), and, in a small percentage of patients, subsequent fibrosis and cirrhosis. In addition, hepatic fat content is closely associated with impaired insulin resistance and type 2 diabetes, conditions increasingly recognized among HIV-infected patients. In the setting of type 2 diabetes mellitus and NASH, thiazolidinediones such as pioglitazone, have been shown to reduce hepatic steatosis, lower transaminase levels and improve insulin sensitivity.

In order to determine the potential benefits of pioglitazone therapy in the setting of HIV infection and hepatic steatosis, we will conduct a 96-week, double-blind, randomized placebo controlled trial of pioglitazone (45 mg/day) in 50 HIV-infected men and women, with 48 weeks of active treatment and 48 weeks of observational follow-up after study treatment ends. We anticipate needing to screen 100 subjects to identify a sufficient number of eligible participants to enroll in the study. The primary outcome variable of interest in this trial will be the change in hepatic fat score, liver-to-spleen ratio, which is calculated from CT scan of the abdomen. Important secondary outcomes will be histologic improvement on liver biopsy performed at baseline and 48 weeks, as well as improvements in transaminase levels and insulin sensitivity measured by hyperinsulinemic euglycemic clamp. All participants will be followed for 48 weeks after discontinuing study treatment to evaluate the short-term natural history of steatosis in those who received placebo and to assess the durability of any potential benefits of pioglitazone upon withdrawal. In this way, important information about the efficacy of pioglitazone to treat hepatic steatosis and improve the metabolic profile in HIV-infected patients will be obtained, as well as preliminary data on whether benefits of pioglitazone are sustained after treatment is discontinued.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Men and women, 18 years of age or greater.
  2. Confirmed HIV infection by ELISA and Western blot.
  3. No changes in antiretroviral regimen within the prior 3 months. Individuals not currently taking antiretroviral therapy will be eligible.
  4. Liver-to-spleen attenuation ratio less than 1 determined by CT and hepatic steatosis on liver biopsy within the past 1 year scored grade 1 or greater (i.e. greater than or equal to 5 percent of hepatocytes).
  5. Fasting glucose less than 126 mg/dL.
  6. Platelets greater than 50,000/microliters.
  7. Willingness to avoid medications and herbal supplements that may increase the risk of bleeding for one week prior to and one week following liver biopsy (e.g. aspirin, NSAIDs and ginko biloba).
  8. Willingness to restrict physical activity 72 hours after liver biopsy.
  9. Willingness to use 2 effective forms of contraception during the study to avoid pregnancy.
  10. Have a primary care physician.

EXCLUSION CRITERIA:

1. Current thiazolidinedione use or use in the last 6 months; known allergy or sensitivity to a thiazolidinedione.
2. Use of insulin or other oral hypoglycemics, or known diabetes.
3. Current pregnancy, breast feeding, or pregnancy within the past 6 months.
4. MELD score greater than 9 or previously diagnosed cirrhosis.
5. ALT greater than 3 times the upper limit of normal.
6. Current or history of heart failure (NYHA Class III or IV cardiac status).
7. Hemoglobin level less than 9g/dL.
8. Active or ongoing infection with Hepatitis A, B, or C.
9. Known or suspected liver disease such as autoimmune hepatitis, Wilson's disease, alpha-1-antitrypsin deficiency, cystic fibrosis, hemachromatosis, glycogen storage disease, amyloidosis, primary biliary cirrhosis, sclerosing cholangitis or any primary or secondary hepatic tumor.
10. Current alcohol/substance abuse or mean alcohol consumption greater than 24g/day over past year.
11. Use of growth hormone, prednisone or other anabolic agents (except for physiologic testosterone replacement) currently or within the past 6 months. One day or less of corticosteroid within the prior 90 days of screening is allowed as is stable dose inhalation corticosteroids.
12. Concurrent use of ketoconazole.
13. Active opportunistic infection (except thrush) or neoplasm (except Kaposi's sarcoma, skin cancer, cancer of the cervix or anus).
14. Any known contraindications to percutaneous liver biopsy including elevated PT/PTT.
15. Severe psychiatric illness that would interfere with adherence to protocol requirements.
16. Known history of insulin secreting tumor or symptomatic hypoglycemia.
17. Current use or a history of treatment with interleukin-2, interferon-alpha, or other investigational agent(s) within the past 6 months. (This does not pertain to ARV's obtained through expanded access).
18. Any medical condition for which the investigator believes a liver biopsy may be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jain MK, Skiest DJ, Cloud JW, Jain CL, Burns D, Berggren RE. Changes in mortality related to human immunodeficiency virus infection: comparative analysis of inpatient deaths in 1995 and in 1999-2000. Clin Infect Dis. 2003 Apr 15;36(8):1030-8. doi: 10.1086/368186. Epub 2003 Apr 2. PMID 12684916
- [Background] Carr A, Samaras K, Chisholm DJ, Cooper DA. Pathogenesis of HIV-1-protease inhibitor-associated peripheral lipodystrophy, hyperlipidaemia, and insulin resistance. Lancet. 1998 Jun 20;351(9119):1881-3. doi: 10.1016/S0140-6736(98)03391-1. PMID 9652687
- [Background] Carr A, Miller J, Law M, Cooper DA. A syndrome of lipoatrophy, lactic acidaemia and liver dysfunction associated with HIV nucleoside analogue therapy: contribution to protease inhibitor-related lipodystrophy syndrome. AIDS. 2000 Feb 18;14(3):F25-32. doi: 10.1097/00002030-200002180-00001. PMID 10716495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment will occur in Clinic 8 of the Clinical Center. We anticipate needing to screen 100 subjects to identify a sufficient number to enroll in the study. Recruitment will be over approximately 1 year.
Groups:
- Placebo: Those participants receiving placebo for 48 weeks
- Pioglitazone 45mg/Day: Those participants receiveing Pioglitazone 45mg/day for 48 weeks.
Period: Overall Study
Arm/Group | Placebo | Pioglitazone 45mg/Day
Started | 25 | 25
Completed | 0 (Study terminated prior to enrollment.) | 0 (Study terminated prior to enrollment.)
Not Completed | 25 | 25
Not completed — Study terminated prior to enrollment | 25 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone 45mg/Day | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 25 | 25 | 50.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 40 (5) | 40 (5) | 40 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25.0
  Male | 13 | 12 | 25.0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50.0

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Steatosis
Description: Evaluation of the safety and potential benefits of pioglitazone therapy on hepatic steatosis in HIV-infected men and women.
Time Frame: 96 weeks
Population: A total of 11 subjects enrolled into the study. 10 were determined to be ineligible during the screening as the Computerized tomography scan revealed a liver-to-spleen ratio > 1 and one was determined ineligible due to concomitant medication use.
Measure: Mean (Standard Deviation); unit: Hounsfeld units
Arm/Group | Placebo | Pioglitazone 45mg/Day
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Insulin Resistance
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Pioglitazone 45mg/Day
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination prior to enrollment leading to no analysis of enrolled participants receiving Pioglitazone or placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes